CLINICAL TRIAL: NCT01433445
Title: A Phase 1b, Open-label, Multi-center, Single Arm, Dose Finding Study to Assess Safety and Pharmacokinetics of the Oral Combination of Panobinostat and Ruxolitinib in Patients With Primary Myelofibrosis (PMF), Post-polycythemia Vera-myelofibrosis (PPV-MF) or Post-essential Thrombocythemia-myelofibrosis (PET-MF)
Brief Title: Panobinostat and Ruxolitinib in Primary Myelofibrosis, Post-polycythemia Vera-myelofibrosis or Post-essential Thrombocythemia-myelofibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589X2106; 2011-000861-10 (EudraCT Number)
Record Dates: First submitted 2011-06-27; First posted 2011-09-14 (Estimated); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Idiopathic Myelofibrosis; Post Essential Thrombocythemia Myelofibrosis; Post Polycythemia-Vera Myelofibrosis
Keywords: Myelofibrosis; Panobinostat; LBH589; Ruxolitinib; MF; PMF; PPV; PPV-MF; PET; PET-MF; JAK2; DACi
MeSH Terms: conditions — Primary Myelofibrosis | interventions — Panobinostat; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): Subjects will be treated with ruxolitinib 5 mg twice daily (BID) and panobinostat 10 mg three times per week (TIW) every other week (QOW) on a 28 day cycle
  Interventions: Drug: panobinostat; Drug: ruxolitinib
- Cohort 2 (Experimental): Subjects will be treated with ruxolitinib 10 mg twice daily (BID) and panobinostat 10 mg three times per week (TIW) every other week (QOW) on a 28 day cycle
  Interventions: Drug: panobinostat; Drug: ruxolitinib
- Cohort 3 (Experimental): Subjects will be treated with ruxolitinib 15 mg twice daily (BID) and panobinostat 10 mg three times per week (TIW) every other week (QOW) on a 28 day cycle
  Interventions: Drug: panobinostat; Drug: ruxolitinib
- Cohort 4 (Experimental): Subjects will be treated with ruxolitinib 15 mg twice daily (BID) and panobinostat 15 mg three times per week (TIW) every other week (QOW) on a 28 day cycle
  Interventions: Drug: panobinostat; Drug: ruxolitinib
- Cohort 5 (Experimental): Subjects will be treated with ruxolitinib 15 mg twice daily (BID) and panobinostat 20 mg three times per week (TIW) every other week (QOW) on a 28 day cycle
  Interventions: Drug: panobinostat; Drug: ruxolitinib
- Cohort 6/6+ (Experimental): Subjects will be treated with ruxolitinib 15 mg twice daily (BID) and panobinostat 25 mg three times per week (TIW) every other week (QOW) on a 28 day cycle
  Interventions: Drug: panobinostat; Drug: ruxolitinib

INTERVENTIONS:
Drug: panobinostat — Given 3 times a week, every other week in 28-day cycles.
  Other Names: LBH589
Drug: ruxolitinib — Given twice daily in 28-day cycles.
  Other Names: INC424

SUMMARY:
This study will assess safety as well as establish a Recommended Phase II dose of the combination of panobinostat and ruxolitinib in patients with or without the JAK2V617F mutation who have been diagnosed with primary myelofibrosis (PMF), Post Essential Thrombocythemia Myelofibrosis (PET MF), or Post-Polycythemia Vera Myelofibrosis (PPV MF).

DETAILED DESCRIPTION:
In 2011 the treatment goals for MF focused on symptom-orientated palliation and quality of life. Both ruxolitinib and panobinostat, as single agents, had shown significant improvement in both of those treatment goals and ruxolitinib had also shown greater reductions in splenomegaly compared to the standard of care at that time. To further the benefit seen with ruxolitinib in MF patients, panobinostat was added to the treatment regimen to act synergistically in the blockade of the dysregulated pathway driving this disease.

The study was conducted in 2 phases - an escalation phase and an expansion phase.

Escalation phase: the study utilised the Bayesian Logistic Regression Model (BLRM), incorporating escalation with overdose control (EWOC), which is a well established method for dose escalation in oncology trials. Following this process, successive cohorts of 3 newly enrolled patients received increasing doses of ruxolitinib and panobinostat until the maximum tolerated dose (MTD) or recommended phase II dose (RPIID) was determined. Once the MTD and/or RPIID were suspected in a minimum of 3 patients, additional patients were enrolled to the same cohort level to reach a minimum of 9 evaluable patients. The process also included safety, PK/PD assessments and estimates of efficacy based on measures of splenic reduction at each dose level.

Expansion: following the determination of the MTD and/or RPIID, a dose expansion phase was conducted at that dose to further define the safety and tolerability of the combination. At least 13, and no more than 23, additional patients were to be enrolled into the expansion phase.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of myelofibrosis, either PMF, PPV or PET MF
* Palpable splenomegaly ≥ 5cm
* May have been previously treated with either panobinostat or ruxolitinib (unless discontinued for clinically relevant toxicities)
* Acceptable lab ranges for all organ systems
* Specifically: Platelet count > 100,000 not reached with the aide of transfusions
* Blast count < 10% at screening
* ECOG ≤ 2
* Must be able to discontinue all drugs being used to treat MF at least 7 days prior to starting study drug

Exclusion Criteria:

* Active malignancy
* Clinically significant heart disease
* Splenic irradiation within 12 months of starting study drug
* Need for ongoing systemic anticoagulation with the exception of Aspirin < 150mg/day or Low Molecular Weight Heparin
* History of platelet dysfunction or bleeding disorder in the 6 months prior to screening
* Patient is at risk for spontaneous bleeding
* Willing and/or eligible for stem-cell transplantation
* Impairment of gastro-intestinal function that may impact the absorption of study treatment
* Unwilling to use highly effective methods of contraception during dosing and for 13 weeks (female participants) or for 6 months (male participants and their female partners) after stopping study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2020-06-22 (Actual); Study Completion 2020-06-22 (Actual)

PRIMARY OUTCOMES:
Rate of dose limiting toxicities at the different dose levels | Cycle 1 (a cycle = 28 days)

SECONDARY OUTCOMES:
Rate of adverse events, serious adverse events, notable laboratory, vital signs and ECG results by dose level | From screening until safety follow up visit (30 days after last treatment), approx. 8.5 years
AUC of ruxolitinib and panobinostat at various dose levels | Ruxolitinib on days 1,2 and 6; Panobinostat on days 2-3 and days 6-7
  Area under the plasma concentration versus time curve
Cmax of ruxolitinib and panobinostat at various dose levels | Ruxolitinib on days 1,2 and 6; Panobinostat on days 2-3 and days 6-7
  Cmax is the Peak Plasma Concentration
Tmax of ruxolitinib and panobinostat at various dose levels | Ruxolitinib on days 1,2 and 6; Panobinostat on days 2-3 and days 6-7
  Tmax: The time of maximum observed concentration sampled during a dosing interval.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- France (2):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Villejuif
- Germany (2):
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
- Ireland (2):
  - Novartis Investigative Site, Dublin
  - Novartis Investigative Site, Galway
- Italy (3):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Varese, VA
- Novartis Investigative Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Novartis Clinical Trials results database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17838